CLINICAL TRIAL: NCT03211208
Title: Assessing Antibiotic Induced Liver Injury for Stratification of Tuberculosis Patients
Acronym: ALISTER
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC16145
Record Dates: First submitted 2017-05-26; First posted 2017-07-07 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Drug-Induced Liver Injury; Anti-Tuberculous Drug Reaction; Tuberculosis
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A panel of highly sensitive circulating biomarkers for acute liver injury have been identified and demonstrated to identify liver injury on first presentation to hospital before standard tests are elevated in patients with paracetamol overdose. The investigators wish to test these biomarkers in patients with active and latent tuberculosis to see if they can be used to stratify patients undertaking anti-tuberculosis drug therapy. Anti-tuberculosis drug induced liver injury is the most frequent side-effect of anti-tuberculosis therapy, affecting 2-5% of tuberculosis patients seen at the Royal Infirmary Edinburgh and hindering their effective treatment. Patients will be recruited from the TB out-patient clinic at the Royal Infirmary Edinburgh. Blood samples will be taken every time the patient visits the clinic and also retrieved from the biochemistry lab. The biomarkers in the blood samples will be analysed to determine if they rise in patients who develop liver injury.

DETAILED DESCRIPTION:
To improve patient stratification, the investigators have developed a panel of novel circulating liver specific and mechanistic biomarkers that report early acute liver injury. Such biomarkers are needed as current early biomarkers of liver injury lack sensitivity and specificity. The panel of biomarkers either have enhanced liver specificity or provide mechanistic insights. Currently, antituberculosis drug-induced liver injury (ATDILI) is the most frequent side-effect of anti-tuberculosis therapy and this hinders the effective treatment of TB, as it means that treatment regimens are not completed. At present, the risk of ATDILI means that monitoring of liver function is required, with levels of ALT measured monthly. If levels of ALT rise to 2-5x the upper limit of normal levels (ULN) and the patient is unwell the frequency of monitoring is increased to biweekly monitoring. Antibiotic therapy is only changed if levels of ALT remain greater than 3xULN, the patient continues to display symptoms and there is a positive causality assessment that the anti-tuberculosis drugs are causing ATDILI. This project will recruit patients taking antituberculosis drugs and determine the diagnostic and prognostic value of the biomarker panel, in relation to liver injury as a result of anti-tuberculosis therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing treatment for tuberculosis
* Patients with the capacity to give consent

Exclusion Criteria:

* Patients unable to give informed consent
* Patients who refuse to take part
* HIV positive patients

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tuberculosis patients being treated at the outpatient clinic at the Royal Infirmary Edinburgh
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
Anti-tuberculosis drug-induced liver injury | Upto 3 years, or until the end of TB treatment
  Anti-tuberculosis drug-induced liver injury defined as ALT elevation more than three times the ULN in the presence of hepatitis symptoms and/or jaundice, or five times the ULN in the absence of symptoms.
  This is a 'proof of concept' study to determine whether a panel of biomarkers are elevated in tuberculosis patients who develop anti-tuberculosis drug-induced liver injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rupprechter SAE, Sloan DJ, Oosthuyzen W, Bachmann TT, Hill AT, Dhaliwal K, Templeton K, Matovu J, Sekaggya-Wiltshire C, Dear JW. MicroRNA-122 and cytokeratin-18 have potential as a biomarkers of drug-induced liver injury in European and African patients on treatment for mycobacterial infection. Br J Clin Pharmacol. 2021 Aug;87(8):3206-3217. doi: 10.1111/bcp.14736. Epub 2021 Jan 26. PMID 33432705